CLINICAL TRIAL: NCT03655288
Title: A Post-marketing Surveillance to Assess Safety and Efficacy of Twotopsplus.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ID-TTP-401
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Post-marketing surveillance of Twotopsplus.

DETAILED DESCRIPTION:
This study will collect clinical data, mainly focused on safety, in Korean population as per the requirement of MFDS for market authorization.

ELIGIBILITY:
Inclusion Criteria:

* The patient diagnosed with hypertension.
* The patient who is first prescribed and administered Twotopsplus Tab.

Exclusion Criteria:

* The patients who are overreacting to this drug or its components.
* The patients with severe renal impairment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient diagnosed with hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-07-25 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse event after this drug administration in general medical practice. | 12weeks
  Any adverse events occurred after this drug dosing will be recorded. Description of adverse event(s) including type of adverse event(s), onset/end date, severity, action taken, causal relationship to the drug and investigator's view on the adverse event(s) will be captured, whether it is related to the drug or not and until follow up visit more than 1 time during the surveillance period.
  Lab abnormalities and changes in vital signs are considered to be adverse events only if they result in discontinuation from the study, necessitate therapeutic medical intervention, and/or if the investigator considers them to be adverse events.
Incidence of serious adverse event after this drug administration in general medical practice | 12weeks
  Any serious adverse events occurred after this drug dosing will be recorded. Description of serious adverse event(s) including type of serious adverse event(s), onset/end date, severity, action taken, causal relationship to the drug and investigator's view on the serious adverse event(s) will be captured, whether it is related to the drug or not and until follow up visit more than 1 time during the surveillance period.
  Lab abnormalities and changes in vital signs are considered to be serious adverse events only if they result in discontinuation from the study, necessitate therapeutic medical intervention, and/or if the investigator considers them to be serious adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea